CLINICAL TRIAL: NCT02329925
Title: The Efficacy of Tongue Stabilizing Device in Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Fernanda Almeida, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H14-01333
Record Dates: First submitted 2014-12-12; First posted 2015-01-01 (Estimated); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tongue Stabilizing Device Treatment (Experimental): Tongue Stabilizing Device (TSD) is a preformed appliance for OSA that protrudes the tongue and improves upper airway structure and function during sleep.
  Interventions: Device: Tongue Stabilizing Device (TSD)

INTERVENTIONS:
Device: Tongue Stabilizing Device (TSD) — Tongue Stabilizing Device (TSD) is a preformed appliance for OSA that protrudes the tongue and improves upper airway structure and function during sleep.

SUMMARY:
The coordination of swallowing and breathing is an important mechanism because the route for air and deglutition is partly shared in the pharynx. Tongue Stabilizing Device (TSD) is a preformed appliance for Obstructive Sleep Apnea (OSA) that protrudes the tongue and improves upper airway structure and function during sleep. Investigators will attempt to assess efficacy of TSD therapy on OSA and the physiological change of swallowing and breathing routes in OSA patients during sleep.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to determine the efficacy of TSD and to assess if it alters swallowing frequency and breathing modes in OSA patients during sleep.

Hypothesis:

Investigators hypothesize that TSD therapy will improve OSA symptoms and will lead to effective nasal breathing which may decrease swallowing frequency in OSA patients during sleep.

Justification:

The coordination of swallowing and breathing is an important mechanism because the route for air and deglutition is partly shared in the pharynx. OSA occurs when there is complete or partial obstruction in the pharynx during sleep which results in an impact on both breathing and swallowing. Continuous Positive Airway Pressure (CPAP) and Oral Appliance (OA) therapy improve breathing in OSA patients, but these therapies have some disadvantages such as poor adherence and expensiveness. TSD is a preformed appliance for OSA that protrudes the tongue and improves upper airway structure and function during sleep. TSD is simpler and more economical than other therapies and may bring similar benefits. In regards to swallowing, it has been reported that swallowing frequency during sleep increases with OSA severity and when preceded by oronasal breathing. However, it still remains to be determined if the treatment of OSA alters breathing modes and swallowing frequency in OSA patients during sleep. An evaluation of the efficacy of TSD therapy on OSA and the physiological change of swallowing and breathing route may be an important step in the sleep medical field so as to understand the mechanism(s) by which TSD therapy improves the clinical condition of OSA.

Objectives:

The objective of this study is to clarify the mechanism(s) by which TSD therapy improves the clinical condition of OSA in terms of regulation of swallowing and breathing modes in OSA patients during sleep.

Research Methods:

Investigators plan to collect data from a minimum of 60 patients who have been diagnosed with OSA .In addition to the regular sleep study electrodes and measurements, investigators will require four supplementary standard sleep channels that utilize standard sleep recording tools. Breathing modes (pure nasal, oral and oro-nasal) will be evaluated with a nasal pressure transducer, which is traditionally used for patients' evaluation (Braebon) and an additional standard oral flow thermistor sensor (1) (Braebon). The degree of mouth opening will be scored with a jaw sensor® (2). Swallowing will be scored based on a combination of measurements which include laryngeal movements as recorded over the thyroid cartilage with a standard piezoelectric sensor (Opti-Flex, Newlife Technologies, Midlothian, VA, USA) (3), and a sub-mental(SupraHyoid) EMG used for the muscle activity of swallowing (4). Standard polysomnography (PSG) data will be analyzed manually according to AASM criteria by sleep technologists. After regular scoring and sleep evaluation, data from results of the sleep study will be transferred to a CD and one of the authors, Kentaro Okuno, will perform further analysis outside of the laboratory. Using the completed data for sleep stages, apnea and hypopnea events, the swallowing events and breathing modes will be assessed visually and scored. Each epoch will then be evaluated for temporal relation between breathing modes and swallowing as well as for degree of mouth opening, apneas, hypopneas, and arousals. The efficacy endpoint is the change in AHI between baseline and TSD. The polysomnographic results will be subjected to paired Student's t-Tests to demonstrate and difference between baseline and TSD.

ELIGIBILITY:
Inclusion Criteria

Patients included in this study must:

* be 18 years of age or older
* have an objective diagnosis of mild to moderate obstructive sleep apnea (OSA) [5 ≤ AHI ≤ 50]; and
* have a Body Mass Index (BMI) ≤ 35

Exclusion Criteria

Patients are excluded in this study who:

* have had previous surgery of the soft palate;
* have neuromuscular disease;
* are taking medications which disturb sleep; and/or
* have ≤ 90% oxygen saturation levels for 20% of the night.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index | At baseline
  Measuring apnea-hypopnea index (events/hour) to measure intervention efficacy (e.g. AHI)
Apnea-hypopnea index | At 2-6 months of TSD treatment follow up
  Measuring changes in apnea-hypopnea index (events/hour) to compare baseline and 2-6 months of TSD treatment follow up.
Frequency of swallowing | At baseline
  Measuring frequency of swallowing (events/hour) to assess influence by intervention
Frequency of swallowing | At 2-6 months of TSD treatment follow up
  Measuring changes in frequency of swallowing (events/hour) to compare baseline and 2-6 months of TSD treatment follow up.

SECONDARY OUTCOMES:
Functional Outcomes of Sleep Questionnaire (FOSQ) responses | At baseline
  Measuring Functional Outcomes of Sleep Questionnaire (FOSQ) responses to evaluate disease specific quality of life.
Functional Outcomes of Sleep Questionnaire (FOSQ) responses | At 2-6 months of TSD treatment follow up
  Measuring changes in Functional Outcomes of Sleep Questionnaire (FOSQ) responses to compare baseline and 2-6 months of TSD treatment follow up
Epworth Sleepiness Scale (ESS) questionnaire responses. | At baseline
  Measuring responses to Epworth Sleepiness Scale (ESS) Questionnaire to assess daytime sleepiness.
Epworth Sleepiness Scale (ESS) questionnaire responses. | At 2-6 months of TSD treatment follow up
  Measuring changes in responses to Epworth Sleepiness Scale (ESS) Questionnaire to compare baseline and 2-6 months of TSD treatment follow up
VR-36 survey responses | At baseline
  Measuring VR-36 survey responses which assesses general health status.
VR-36 survey responses | At 2-6 months of TSD treatment follow up
  Measuring changes in VR-36 survey responses to compare baseline and 2-6 months of TSD treatment follow up
Breathing route | At baseline
  Measuring breathing route to assess influence by intervention
Breathing route | At 2-6 months of TSD treatment follow up
  Measuring changes in breathing route to compare baseline and 2-6 months of TSD treatment follow up
Swallowing apnea time | At baseline
  Measuring swallowing apnea time (sec) to assess influence by intervention
Swallowing apnea time | At 2-6 months of TSD treatment follow up
  Measuring changes in swallowing apnea time (sec) to compare baseline and 2-6 months of TSD treatment follow up
Compliance (Measuring adherence (hours/nights and nights/week of intervention use)) | At 2-6 months of TSD treatment follow up
  Measuring adherence (hours/nights and nights/week of intervention use)

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda R Almeida, DDS, MSc, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Alshhrani WM, Hamoda MM, Okuno K, Kohzuka Y, Fleetham JA, Ayas NT, Comey R, Almeida FR. The efficacy of a titrated tongue-stabilizing device on obstructive sleep apnea: a quasi-experimental study. J Clin Sleep Med. 2021 Aug 1;17(8):1607-1618. doi: 10.5664/jcsm.9260. PMID 33745505